CLINICAL TRIAL: NCT04913103
Title: A Phase II, Open-label Study of Polatuzumab-vedotin (PV) in Combination With Bendamustine and Rituximab for Patients With Mantle Cell Lymphoma, Who Relapse After Previous Therapy With Bruton Tyrosine Kinase Inhibitor
Brief Title: Study of PV in Combination With Bendamustine and Rituximab for Patients With R/R MCL
Acronym: CLSGMCLPOLA
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Czech Lymphoma Study Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLSG-MCL-POLA
Record Dates: First submitted 2021-05-19; First posted 2021-06-04 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-05

CONDITIONS: Lymphoma, Mantle-Cell
Keywords: refractory/relapsed mantle cell lymphoma; polatuzumab-vedotin; bendamustine; rituximab
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — polatuzumab vedotin; Bendamustine Hydrochloride; Rituximab

STUDY DESIGN:
Intervention Model Description: open-label, single arm, combination - polatuzumab vedotine + rituximab+bendamustin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm, open-label (Experimental): combination of polatuzumab-vedotin, bendamustine and rituximab
  Interventions: Drug: Polatuzumab vedotin; Drug: Bendamustine Hydrochloride; Drug: Rituximab

INTERVENTIONS:
Drug: Polatuzumab vedotin — treatment by a study drug polatuzumab-vedotin, i.v.
  Other Names: Polivy
Drug: Bendamustine Hydrochloride — treatment by a study drug bendamustin i.v.
  Other Names: Bendamustine Accord; Bendamustine Glenmark; Bendamustine KABI
Drug: Rituximab — treatment by a study drug rituximab, i.v.
  Other Names: Mabthera; Rixathon; Truxima

SUMMARY:
A Czech Lymphoma Study Group, phase II, open-label, study of polatuzumab-vedotin in combination with bendamustine and rituximab for patients with mantle cell lymphoma, who relapse after previous therapy with Bruton tyrosine kinase inhibitor

DETAILED DESCRIPTION:
Primary objective:

Efficacy: to evaluate the efficacy of the combination of polatuzumab vedotin plus bendamustine and rituximab (BR) with respect to progression-free survival (PFS)

Secondary objectives:

Efficacy: to evaluate the efficacy of polatuzumab vedotin plus BR with respect to secondary efficacy endpoints, namely overall response rate, duration of response, event free survival and overall survival; Safety objective; Exploratory objectives

ELIGIBILITY:
Inclusion Criteria:

* Signed written Informed Consent Form
* Adult patients with relapsed or refractory MCL after failure of BTK inhibitor-containing therapy (e.g. ibrutinib, acalabrutinib, zanubrutinib)
* Patients previously treated with bendamustine are eligible for the study treatment, in the case they had achieved objective response (CR or PR) and the last dose of bendamustine was administered ≥ 1 year before the estimated study treatment initiation date (C1D1)
* Tumor tissue at the lymphoma relapse after failure of BTK inhibitor. In case that a re-biopsy is not possible (e.g. urgent need to start study treatment), archival tissue blocks may be used to confirm the diagnosis
* Bone marrow examination by standard trephine biopsy including flow cytometry analysis within 8 weeks before study entry
* Age 18-80 years at the time of signing Informed Consent Form
* ECOG Performance Status of 0, 1, or 2
* Life expectancy ≥ 2 months
* Adequate hematologic function (unless due to underlying disease, as established for example, by extensive bone marrow involvement or due to hypersplenism secondary to the involvement of the spleen by MCL per the investigator), defined as follows:

  * Hemoglobin ≥ 80g/L
  * ANC ≥ 1,500/μL
  * Platelet count ≥ 75,000/μL Enrollment of patients with lower counts is possible only after consulting the medical monitor.
* Adequate cardiac functions according to echocardiography (ECHO) within 6 months before study entry
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for at least 12 months after the last dose of study treatment. Women must refrain from donating eggs during this same period. A woman is considered to be of childbearing potential if she is post-menarcheal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus). The definition of childbearing potential may be adapted for alignment with local guidelines or requirements.

Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.

The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or post-ovulation methods) and withdrawal are not acceptable methods of contraception.

* For women of childbearing potential, a negative serum pregnancy test result within 7 days prior to commencement of dosing. Women who are considered not to be of childbearing potential are not required to have a pregnancy test.
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm, as defined below:

With female partners of childbearing potential or pregnant female partners, men must remain abstinent or use a condom during the treatment period and for at least 5 months after the last dose of polatuzumab vedotin, 3 months after the last dose of rituximab, and for at least 6 months after the last dose of bendamustine to avoid exposing the embryo for the duration of the pregnancy. Men must refrain from donating sperm during this same period. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of preventing drug exposure. Male patients considering preservation of fertility should bank sperm before study treatment.

Exclusion Criteria:

* Prior organ transplantation
* Current Grade ≥ 2 peripheral neuropathy by clinical examination or demyelinating form of Charcot-Marie-Tooth disease
* History of other malignancy that could affect compliance with the protocol or interpretation of results Patients with a history of curatively treated basal or squamous cell carcinoma or melanoma of the skin or in situ carcinoma of the cervix at any time prior to the study are eligible Patients with any malignancy appropriately treated with curative intent and the malignancy has been in remission without treatment for ≥ 2 years prior to enrollment are eligible Patients with low-grade, early-stage prostate cancer (Gleason score 6 or below, Stage

  1 or 2) with no requirement for therapy at any time prior to study are eligible.
* Evidence of significant, uncontrolled, concomitant diseases that could affect compliance with the protocol or interpretation of results.
* Recent major surgery (e.g. within 4 weeks prior to the start of Cycle 1), other than for diagnosis
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment or significant infections within 2 weeks before the start of Cycle 1.
* Clinically significant liver disease, including active viral or other hepatitis, current alcohol abuse, or cirrhosis
* Illicit drug or alcohol abuse within 12 months prior to screening, in the investigator's judgment
* Any of the following abnormal laboratory values (unless any of these abnormalities are due to underlying lymphoma):

INR > 1.5 x upper limit of normal (ULN) in the absence of therapeutic anticoagulation aPTT > 1.5 x ULN in the absence of a lupus anticoagulant

* Serum AST and ALT > 3 x ULN
* Total bilirubin > 2 x ULN Patients with documented Gilbert disease may be enrolled if total bilirubin is > 3.0 x ULN.
* Serum creatinine clearance < 40 mL/min (using Cockcroft-Gault formula or creatinine levels assessed directly from the collected urine)
* Patients with suspected active or latent tuberculosis (as confirmed by a positive interferon-gamma release assay)
* Positive test results for chronic hepatitis B infection defined as positive hepatitis B surface antigen (HBsAg) serology
* Patients with occult or prior hepatitis B infection defined as positive total hepatitis B core antibody and negative HBsAg may be included if hepatitis B virus (HBV) DNA is undetectable at the time of screening. These patients must be willing to undergo regular DNA testing and appropriate antiviral therapy as indicated.
* Positive test results for hepatitis C virus (HCV) antibody serology testing Patients positive for HCV antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
* Known history of HIV seropositive status
* Patients with a history of progressive multifocal leukoencephalopathy
* Pregnancy or lactation or intending to become pregnant during study
* CNS lymphoma In patients with clinical signs attributable to CNS lymphoma, CT scan (MRI also acceptable) of the head and examination of cerebrospinal fluid will be required prior to study treatment initiation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 4 years
  evaluation of the efficacy of the combination of polatuzumab vedotin plus bendamustine and rituximab (BR) with respect to progression-free survival (PFS)

SECONDARY OUTCOMES:
overall response rate (ORR) | 4 years
  efficacy of polatuzumab vedotin plus BR with respect to overall response rate
duration of response (DoR) | 4 years
  efficacy of PV plus BR with respect to duration of response
event free survival (EFS) | 4 years
  efficacy of PV plus BR with respect to event free survival
overall survival (OS) | 4 years
  efficacy of PV plus BR with respect to overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Klener, Prof.MD,PhD, Principal Investigator — Czech Lymphoma Study Group
Locations (7):
- Czechia (7):
  - University Hospital Brno, Brno
  - University Hospital Hradec Králové, Hradec Králové
  - University Hospital Olomouc, Olomouc
  - University Hospital Ostrava, Ostrava
  - University Hospital Plzeň, Pilsen
  - University Hospital Kralovske Vinohrady, Prague
  - Charles University General Hospital, Prague

IPD SHARING:
Plan to Share IPD: No